CLINICAL TRIAL: NCT03948607
Title: Neural Mechanisms Underlying Attention Lapses in Adult Attention Deficit Disorder: Towards a Better Clinical Diagnosis
Brief Title: Neural Mechanisms of Attention Lapses in Adult ADHD
Acronym: AttLapse-TDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7248
Record Dates: First submitted 2019-03-11; First posted 2019-05-14 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Attention Deficit Disorder; Hyperactivity Disorder
Keywords: Electroencephalography; Neurocognition; Attention deficit; Attention lapses
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult ADHD: Adult ADHD patients without current comorbidity and treatment.
  Interventions: Other: Electroencephalography during sustained attention task.
- Healthy controls: Healthy controls without ADH, paired in age and gender.
  Interventions: Other: Electroencephalography during sustained attention task.

INTERVENTIONS:
Other: Electroencephalography during sustained attention task. — The Continuous Temporal Expectancy Task (CTET) (O'Connell et al., 2009) is a very demanding discrimination task with sustained attention. It consists of the presentation on a computer screen of a visual pattern resembling a checkerboard that changes orientation at regular intervals of time. In this task the subject must respond (pressing a response button) to the appearance of rare target stimuli that have a longer duration (1120 ms) than non-target stimuli (800 ms).
  SART (Sustained Attention to Response Task) (Robertson et al., 1997) is a task of inhibition (Go / No-Go task) to evaluate the capacities of sustained attention. It consists in the successive and random presentation on a computer screen of the numbers from 1 to 9. In this task the subject must respond, by pressing a response button, to the appearance of all the numbers (very non-target stimuli frequent), with the exception of the number "3".
  Other Names: CTET (Continuous Temporal Expectancy Task); SART (Sustained Attention to Response Task)

SUMMARY:
ADHD is a common disorder, leading to a significant disability that often persists in adulthood. ADHD is characterized by attentional disturbances that are difficult to asses with standard neuropsychological tests.

Attention tends to stall after a certain time of fatigue (i.e. an attention lapse). The aim of this study is to study the electroencephalographic (EEG) characteristics of these attention lapses in a sustained attention task, comparing ADHD patients with healthy subjects.

DETAILED DESCRIPTION:
The main goal is to assess with EEG the timing of the attentional demobilization that precedes a sustained attention lapse in patients with ADHD.

The secondary objectives are: 1 / To analyze impaired cognitive control mechanisms during lapses in patients with ADHD; 2 / Study the relationships between the deficits identified through EEG recording, clinical evaluations, and the subjective perception of daily difficulties; 3 / To measure the impact of the subjective attention state on the neuronal precursors of the attentional lapses; 4 / Evaluate the relation between propensity to wandering mind and attentional lapses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD according to DSM-5 criteria by a psychiatrist with clinical experience with ADHD
* aged 18 to 60
* having signed an informed consent
* able to understand the objectives and the risks related to the research

For Healthy controls

* Absence of psychiatric disorder or neurological disease
* Matched in sex, age (± 2 years) and level of study (± 2 years) to each ADHD patient

Exclusion criteria:

* treatment by Methylphenidate or amphetamine in the 3 months preceding the study
* treatment by a psychotropic drug other than antidepressant SSRI: anti-depressant non-SSRI, antipsychotic, mood stabilizer, benzodiazepine or hypnotic daily intake
* neurological pathology or neurological sequelae
* history of head trauma with loss of consciousness of more than 15 minutes
* Subject under the protection of justice
* Subject under guardianship, curatorship
* Subject in exclusion period (determined by previous or current study),
* Impossibility to give the subject enlightened information (subject in emergency situation, difficulties of comprehension of the subject (for example mental retardation, illiteracy, subject not including French ...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients included in the ADHD group are patients assessed during a specialized consultation on adult ADHD This consultation corresponds to standard care, during which a clinical examination is performed, as well as an interview with the psychiatrist.
  If the diagnosis of ADHD is confirmed, comorbidities are systematically sought and the eligibility criteria for inclusion of the patient in the study are verified.
  Healthy control are recruited by advertising.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Spectral amplitude of the alpha band (8-14 Hz) to the quantitative EEG during the period up to 20 seconds before the successful trials vs. missed trials (lapse). | During EEG realized after the inclusion
  In healthy subjects, EEG changes, including increased parieto-occipital activity in the alphas frequency band (8-14Hz), have been observed 20 seconds before lapse (O'Connell et al., 2009). The analysis of the evoked potentials associated with the stimuli presented just before the occurrence of the target stimulus, reveals that the amplitude of the P300 on the 5 trials preceding the target to be detected is significantly lower before an omission (lapse) than before a correct detection.

SECONDARY OUTCOMES:
CNV difference between missed and successful trials | During EEG realized after the inclusion
  Time course analysis of electrophysiological markers (EEG) before an attention lapse : amplitude of the evoked potentials
CNV difference between missed and successful trials | During EEG realized after the inclusion
  Time course analysis of electrophysiological markers (EEG) after a successful test: amplitude of the evoked potentials and theta power (intensity in μV).
Association between EEG lapses markers, neuropsychological measures of attention, clinical scales and subjective mindwandering | During EEG realized after the inclusion
  Regression and correlation analyzes involving electrophysiological markers associated with attentional lapses (see main objective)
Association between EEG lapses markers, neuropsychological measures of attention, clinical scales and subjective mindwandering | During EEG realized after the inclusion
  Regression and correlation analyzes involving electrophysiological markers associated with neuropsychological attention test scores (TAP)
Association between EEG lapses markers, neuropsychological measures of attention, clinical scales and subjective mindwandering | During EEG realized after the inclusion
  Regression and correlation analyzes involving electrophysiological markers associated with clinical scales (self-report ASRS and WFIRS)
Association between EEG lapses markers, neuropsychological measures of attention, clinical scales and subjective mindwandering | During EEG realized after the inclusion
  Regression and correlation analyzes involving electrophysiological markers associated with subjective measures of mind wandering (ad hoc questionnaire)
EEG lapse markers according attentional subjective state | During EEG realized after the inclusion
  Frequency of lapses of attentional lapses (evoked potentials P3a and CNV, theta power) (intensity in μV), according to the attentional state described by the subjects during the evaluations during the task
EEG lapse markers according attentional subjective state | During EEG realized after the inclusion
  amplitude electrophysiological markers (EEG) of attentional lapses (evoked potentials P3a and CNV, theta power) (intensity in μV), according to the attentional state described by the subjects during the evaluations during the task

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien WEIBEL, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpital Civil - service de Psychiatrie 2, Strasbourg, France